CLINICAL TRIAL: NCT04057196
Title: Self-System Therapy for Older Adults With Advanced Lung Cancer (SST-LC)
Brief Title: Self-System Therapy for Older Adults With Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00102705
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer Stage III; Lung Cancer Stage IV
MeSH Terms: conditions — Lung Neoplasms | interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with Advanced Lung Cancer (Experimental): Older adults with stage III or stage IV lung cancer will be enrolled in the Self-System Therapy intervention to treat illness-related distress, depression, and to enhance self-efficacy via delivery of behavioral coping skills across a period of 12 weeks.
  Interventions: Behavioral: Self-System Therapy for Older Adults with Advanced Lung Cancer (SST-LC)

INTERVENTIONS:
Behavioral: Self-System Therapy for Older Adults with Advanced Lung Cancer (SST-LC) — The SST-LC is a brief structured intervention deliverable by video conference. The new SST-LC protocol will incorporate behavioral strategies designed to meet the needs of older adults with lung cancer, including examining individual and shared expectations for lung cancer care, identifying discrepancies between expectations and realistic possibilities, and modifying stress-exacerbating behaviors.

SUMMARY:
The purpose of this study to use Self-system therapy (SST), to treat depression and lung-cancer-related distress in older adults (65 years and older).

DETAILED DESCRIPTION:
The investigator will examine whether delivering the SST intervention will be both feasible and acceptable to study participants. The investigator will also examine whether participation in SST can help alleviate symptoms of depression and distress while helping improve overall functioning in older adults with advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* English-speaking
* The patient has a diagnosis of late-stage (III-IV) lung cancer and is living at her/his home.

Exclusion Criteria:

* Unable to provide informed consent
* Visual or hearing impairments that preclude participation
* Serious mental illness

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Ramos, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strauman TJ, Eddington KM. Treatment of Depression From a Self-Regulation Perspective: Basic Concepts and Applied Strategies in Self-System Therapy. Cognit Ther Res. 2017 Feb;41(1):1-15. doi: 10.1007/s10608-016-9801-1. Epub 2016 Aug 29. PMID 28216800
- [Background] Waters SJ, Strauman TJ, McKee DC, Campbell LC, Shelby RA, Dixon KE, Fras AM, Keefe FJ. Self-system therapy for distress associated with persistent low back pain: A randomized clinical trial. Psychother Res. 2016 Jul;26(4):472-83. doi: 10.1080/10503307.2015.1040485. Epub 2015 Jun 16. PMID 26079438
- [Derived] Ramos K, Ayaz A, Riley J, Faircloth K, Porter LS, Strauman TJ. Adaptation and Implementation of Self-System Therapy for Older Adults with Advanced Lung Cancer: Pilot Trial Results. Cancers (Basel). 2025 Aug 28;17(17):2809. doi: 10.3390/cancers17172809. PMID 40940906

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adults With Advanced Lung Cancer
Started | 30
Completed | 24
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.77 (4.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Complete SST Treatment Sessions
Description: Completion of at least 85% of SST treatment sessions across a 12-week period.
Time Frame: up to week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
Participants | 23

2. Primary Outcome: Patient Satisfaction With Treatment
Description: The Client Satisfaction Questionnaire (CSQ-8), which assesses treatment credibility (pre-treatment) and effectiveness of/satisfaction with services (post-treatment). An overall score is calculated by summing the respondent's rating (item rating) score for each scale item. For the CSQ-8 version, scores therefore range from 8 to 32, with higher values indicating higher satisfaction.
Time Frame: End of study, week 12
Population: Data not collected on 7 participants (3 withdrew prior to the study, 3 completed less than 8 sessions, and one who died from their lung cancer and could not complete).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 23
score on a scale | 30.78 (1.78)

3. Secondary Outcome: General Distress as Measured by the CORE-10 (Clinical Outcomes in Routine Evaluation 10) at Baseline
Description: The CORE-10 measure will be used for rating general distress. The measure comprises ten questions about how participants have been feeling over the past week. Scores range from 0-40, with higher scores indicating greater distress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
score on a scale | 14.55 (3.93)

4. Secondary Outcome: General Distress as Measured by the CORE-10 at 12 Weeks
Description: as for outcome 3
Time Frame: 12 weeks
Population: Seven participants had been withdrawn from the study at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 23
score on a scale | 12.67 (3.62)

5. Secondary Outcome: General Distress as Measured by the CORE-10 at 1-month Follow-up
Description: as for outcome 3
Time Frame: 1-month follow-up, up to 4 months
Population: Nine participants did not complete due to withdrawal or death.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 21
score on a scale | 12.30 (3.60)

6. Secondary Outcome: Depression as Measured by the Beck Depression Inventory (BDI-II) at Baseline
Description: Depression will be measured using the Beck Depression Inventory (BDI-II). The measure has 21 items. The BDI-II is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The total score ranges from 0 to 63, where higher scores indicate greater depression.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
score on a scale | 9.41 (6.09)

7. Secondary Outcome: Depression as Measured by the Beck Depression Inventory (BDI-II) at 12 Weeks
Description: as for outcome 6
Time Frame: 12 weeks
Population: Seven participants had been withdrawn from the study at 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 23
score on a scale | 6.17 (6.07)

8. Secondary Outcome: Depression as Measured by the Beck Depression Inventory (BDI-II) at 1-month Follow-up
Description: as for outcome 6
Time Frame: 1-month follow-up, up to 4 months
Population: Nine participants did not complete due to withdrawal or death.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 21
score on a scale | 6.13 (5.10)

9. Secondary Outcome: Functioning as Measured by the Functional Assessment of Cancer Therapy- Lung (FACT-L)
Description: Functioning will be measured using the Functional Assessment of Cancer Therapy- Lung (FACT-L). The FACT-L is a 36-item measure, each item with a five-point scale from 0 (not at all) to 4 (very much), measuring overall quality of life (QOL) across five dimensions that are summed together to derive a total score. The total score range is from 0-136. The higher the score, the better the QOL.
Time Frame: Baseline, 12 weeks, 1 month follow-up (up to 4 months)
Population: Participants with FACT-L scores available at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
score on a scale
  Baseline | 102.22 (16.71)
  12 weeks: number analyzed (Participants) | 23
  12 weeks | 109.12 (16.01)
  1 month follow-up: number analyzed (Participants) | 21
  1 month follow-up | 101.47 (17.51)

10. Secondary Outcome: Number of Participants With Participant-reported Mobility Indices Available
Description: Mobility indices will include participant report of difficulty walking across a room without help from another person or equipment (none, a little vs some, a lot, unable), difficulty walking two to three blocks without help from another person or equipment (none, a little vs some, a lot, unable), and use of assistive device (yes vs no).
Time Frame: Baseline, 12 weeks, 1 month follow-up (up to 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
Participants
  Baseline | 30
  12 weeks | 23
  1 month follow-up | 21

11. Secondary Outcome: Number of Participants With Physical Activity Scale for the Elderly (PASE) Scores Available
Description: Physical Activity will be measured using the Physical Activity Scale for the Elderly (PASE)The instrument is comprised of self-reported occupational, household and leisure activities items over a one-week period. PASE scores are calculated from weights and frequency values for each of 12 types of activity.
Time Frame: Baseline, 12 weeks, 1 month follow-up (up to 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
Participants
  Baseline | 30
  12 weeks | 23
  1 month follow-up | 21

12. Secondary Outcome: Number of Participants With Computerized Selves Questionnaire (CSQ) Responses Available at Baseline
Description: Self-Discrepancy will be measured using the Computerized Selves Questionnaire (CSQ). The CSQ is a computer-based version of the original self-discrepancy questionnaire used by Higgins and colleagues (1986) in which a person is asked to produce a list of eight personal attributes that s/he would ideally like to possess and eight attributes s/he feels s/he ought to possess. To score, qualities in the actual self column are compared with those in the ought self column.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
Participants | 30

13. Secondary Outcome: Number of Participants With Regulatory Focus Questionnaire (RFQ) Responses Available at Baseline
Description: Self-Regulatory Orientation will be measured using the Regulatory Focus Questionnaire (RFQ).The measure has 11 items using 5-point scales, along two sub scales measuring the extent to which an individual believes s/he has been successful in attaining promotion or prevention goals. Six questions quantify Promotion and five questions quantify Prevention the promotion sums must be divided by 6, and the prevention sums must be divided by 5 in order to place scores for both orientations on the same 1-5 scale.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
Participants | 30

14. Secondary Outcome: Treatment Session Fidelity as Measured by Number of Participants Who Were Taught All Skills.
Description: Trained raters will listen to audio recordings of treatment sessions and use a pre-defined checklist of session content and strategies of the treatment to indicate if session coping skills were taught (yes/no) coded as 1 for yes and 0 for no. Higher scores indicate greater session fidelity.
Time Frame: End of study, week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 30
Participants | 24

ADVERSE EVENTS:
Time Frame: At 12 weeks and 1-month follow-up.
Description: Reporting of patients with late-stage lung cancer who died due to progressing illness, not linked to participation in SST-LC behavioral intervention.
Arm/Group | Adults With Advanced Lung Cancer
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults With Advanced Lung Cancer (N=30)
Unfavorable changes in health, due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT04057196/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT04057196/ICF_000.pdf